CLINICAL TRIAL: NCT03046251
Title: Natalizumab in Preventing Post-partum Relapses in Multiple Sclerosis
Acronym: NAPPREMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Bianca Weinstock-Guttman, Professor of Neurology, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: US-TYS-14-10720
Record Dates: First submitted 2017-02-03; First posted 2017-02-08 (Estimated); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- natalizumab (Other): Participants in this group are those who opt to receive treatment with natalizumab IV 300mg/day given q 4 weeks for 48 weeks.
  Interventions: Drug: Natalizumab
- Control (No Intervention): Participants in this group may initiate any FDA approved DMT at any time post delivery or remain on no therapy.

INTERVENTIONS:
Drug: Natalizumab
  Arms: natalizumab

SUMMARY:
The purpose of this study is to evaluate if monthly natalizumab, initiated after delivery, is effective in preventing postpartum relapses.

DETAILED DESCRIPTION:
Postpartum patients with a diagnosis of multiple sclerosis (MS) will be given the opportunity to enroll in this study that will evaluate the efficacy of IV natalizumab to prevent postpartum relapses. Natalizumab, administered as 300mg IV q 4 weeks, will be initiated postpartum (0-30 days post-delivery).

Patients who decline natalizumab treatment postpartum will be given the opportunity to enroll in the study in the control group. The control group will have similar inclusion and exclusion criteria as well as scheduled visit and study procedures as the active natalizumab treatment group.

The primary objective of the trial is to assess the efficacy of IV administered natalizumab, monthly for 1 year, in preventing relapses during the postpartum period.

The secondary objectives of the trial are to assess the efficacy of natalizumab in decreasing the risk for disability progression during the postpartum period and to prevent the appearance of new and/or enlarging brain MRI lesions as measured by qualitative MRI analysis.

The tertiary objective is to assess the association of the clinical outcomes with subject evaluations including patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects postpartum, 0-30 days postpartum at the time of informed consent.
2. Diagnosis of relapsing form of MS.
3. Willing to initiating natalizumab and enroll in the TOUCH system.
4. Willing and able to comply with the study procedures for the duration of the trial.
5. Signed informed consent and HIPAA authorization.

Exclusion Criteria:

1. Diagnosis of primary progressive MS.
2. Breastfeeding
3. Use of IVIG in Tysabri treated subjects.
4. Significant renal or hepatic impairment (in the opinion of the investigator) or other significant disease (e.g., cognitive impairment) that would compromise adherence and completion of the trial.
5. History of hypersensitivity to previous exposure or presence of antibodies to natalizumab.
6. Any other factor that, in the opinion of the investigator, would make the subject unsuitable for participation in this study.
7. Patients that experience relapses and/or initiated DMT's during pregnancy

The Control group will consist of relapsing MS patients post-delivery who decline natalizumab therapy but open to enroll in the study.

Similar Inclusion and Exclusion criteria as the natalizumab group with the exception of requiring TOUCH enrollment program. The Control group will be allowed to initiate any FDA approved DMT at any time post delivery or remain on no therapy while breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Weinstock-Guttman, MD, Principal Investigator — SUNY Buffalo
Locations (1):
- SUNY Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Post-delivery patients enrolled and followed for 52 weeks. Study had difficulty in enrollment locally (Buffalo).
Groups:
- Natalizumab: Participants in this group are those who opt to receive treatment with natalizumab IV 300mg/day given q 4 weeks for 48 weeks.
  Natalizumab
Period: Overall Study
Arm/Group | Natalizumab | Control
Started | 4 (Post-delivery start after 4 weeks) | 26
Completed | 4 (Monitored for 52 weeks post-delivery) | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 30 patients enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Natalizumab | Control | Total
Number analyzed (Participants) | 4 | 26 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (4.3) | 31.8 (5.6) | 32.3 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 26 | 30
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 3 | 22 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 26 | 30
Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: units on a scale] — The Expanded Disability Status Scale (EDSS) is a measure used to assess disability levels in individuals with multiple sclerosis. It ranges from 0 (no disability) to 10 (death due to MS). Scores from 1.0 to 4.5 indicate patients with significant ambulatory abilities, while scores from 5.0 to 9.5 reflect progressive loss of mobility.
  units on a scale | 2.0 (0.0) | 1.5 (0.9) | 1.6 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Relapses Post Partum
Description: The primary endpoint are the relapses during 1 year post-delivery in patients treated with natalizumab. This will be compared to the relapse frequency in the parallel control group.
Time Frame: 52 weeks
Population: Two of the 4 natalizumab users reported post-partum relapses, compared to 7 out of the 24 who were not using natalizumab post-partum.
Measure: Count of Participants; unit: Participants
Arm/Group | Natalizumab | Control
Number analyzed (Participants) | 4 | 24
Participants | 2 | 7

2. Secondary Outcome: Expanded Disability Status Scale (EDSS) Worsening
Description: EDSS scores were determined at multiple timepoints, with scores nearest to week 52 selected for analysis. The difference between EDSS scores at baseline and week 52 were calculated, categorizing patients into two groups: stable or worsened. EDSS worsening was defined as a 1.0 increase for baseline scores below 6.0, or a 0.5-point increase for baseline scores of 6.0 or higher.
Time Frame: 52 weeks
Population: Number of patients who worsened in EDSS scores comparing baseline visit to visit closest to 52 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Natalizumab | Control
Number analyzed (Participants) | 3 | 25
Participants | 0 | 4

3. Secondary Outcome: Difference in Mean Expanded Disability Status Scale (EDSS) Scores Between Persons With MS (pwMS) Treated With Natalizumab Versus Other Disease-modifying Therapies (DMT)
Description: The Expanded Disability Status Scale (EDSS) is a standardized measure of disability progression in multiple sclerosis (MS), ranging from 0 to 10 in 0.5-unit increments, with higher scores indicating greater disability. EDSS scores were determined at multiple timepoints, with scores nearest to week 52 selected for analysis.
Time Frame: 52 weeks
Population: Persons with MS with available EDSS scores comparing the visit closest to 52 weeks between those treated with natalizumab vs other DMTs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Natalizumab | Control
Number analyzed (Participants) | 4 | 25
score on a scale | 1.8 (0.5) | 1.8 (1.0)

4. Secondary Outcome: Change in MRI
Description: The patients with MS (pwMS) underwent at least two MRI examinations: the first occurring 1-3 months postpartum (before the first post-partum dose of natalizumab) and a follow-up MRI closest to the week 52 visit. For this study, T2-FLAIR and T1-weighted sequences were acquired before and after gadolinium contrast administration. A licensed and experienced neuroradiologist analyzed the MRI scans, determining the number of new or newly enlarging T2 lesions and new T1 contrast-enhancing (GdE) lesions. The identification of new lesions was based on comparisons with pre-pregnancy scans.
Time Frame: 52 weeks
Population: Patients with MS (pwMS) with available MRI data
Measure: Count of Participants; unit: Participants
Arm/Group | Natalizumab | Control
Number analyzed (Participants) | 4 | 18
Participants
  New T2 lesions | 3 | 5
  NEW GdE lesions: number analyzed (Participants) | 4 | 17
  NEW GdE lesions | 1 | 3

5. Secondary Outcome: Percent of Relapse Free Patients
Description: Percent of relapse free patients between the groups
Time Frame: 52 weeks
Population: Relapse free at 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Natalizumab | Control
Number analyzed (Participants) | 4 | 24
Participants | 2 | 17

6. Other Pre Specified Outcome: Change in QoL Measures
Description: The study participants completed multiple patient-reported outcome (PRO) questionnaires: the Multiple Sclerosis Impact Scale-29 (MSIS-29) and the Fatigue Scale for Motor and Cognitive Function (FSMC). The MSIS-29 is a psychometrically validated 29-item measure widely used in MS treatment trials, consisting of two domains: a 20-item physical impact subscale and a 9-item psychological impact subscale. The FSMC is a 20-item scale designed to assess fatigue in MS patients, with 10 items each for cognitive and motor fatigue. Both scales have proven to be valuable tools in assessing the impact of MS on patients' daily lives and are frequently used in clinical trials and research settings.
Time Frame: 52 weeks
Population: Worsening of MSIS physical, mental, or FSMC worsening comparing baseline to week 52.
Measure: Count of Participants; unit: Participants
Arm/Group | Natalizumab | Control
Number analyzed (Participants) | 4 | 18
Participants
  MSIS Physical Worsening | 3 | 9
  MSIS Mental Worsening | 4 | 9
  FSMC Worsening | 4 | 9

7. Other Pre Specified Outcome: Proportion of Postpartum MS Patients With Disability Progression Comparing Those Who Used a Disease Modifying Therapy (DMT) After Delivery vs Those Who Did Not Re-start a DMT After Delivery.
Description: To evaluate the impact of postpartum DMT use on disability progression, we compared the proportion of patients experiencing confirmed EDSS worsening at 52 weeks between those who restarted DMT after delivery and those who did not. Confirmed EDSS worsening was defined as an increase of ≥1.0 point from baseline for patients with baseline EDSS <6.0, or ≥0.5 points for patients with baseline EDSS ≥6.0, sustained for at least 12 weeks.
Time Frame: 52 weeks
Population: Persons with MS (pwMS) who participated in this study.
Measure: Count of Participants; unit: Participants
Groups:
- DMT Used: DMT restarted within 1 year postpartum
- No DMT Used: DMT not restarted within 1 year postpartum
Arm/Group | DMT Used | No DMT Used
Number analyzed (Participants) | 22 | 6
Participants | 3 | 1

8. Other Pre Specified Outcome: Difference in EDSS Scores Between Patients With MS (pwMS) Who Used a Disease Modifying Therapy (DMT) After Delivery vs Those Who Did Not Re-start a DMT After Delivery.
Description: To evaluate the impact of postpartum DMT use on disability progression, we compared the mean EDSS scores (a standardized measure of MS disability ranging from 0-10) at 52 weeks between patients who restarted DMT after delivery and those who did not.
Time Frame: 52 weeks
Population: Persons with MS (pwMS) who participated in this study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DMT Used | No DMT Used
Number analyzed (Participants) | 23 | 6
score on a scale | 1.7 (0.8) | 2.3 (1.2)

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Serious side effects Infections Jaundice Anemia Allergy or infection in the brain Acute hypersensitivity reactions Cholelithiasis
  Common side effects Headache Fatigue Urinary tract infection Joint pain Lung infection Depression Pain in arms or legs Diarrhea Vaginitis Rash Relapse not requiring hospitalization
Arm/Group | Natalizumab | Control
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/26
Other Adverse Events (participants affected / at risk) | 2/4 | 7/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natalizumab (N=4) | Control (N=26)
MS relapse (Nervous system disorders) | 2 (2) | 7 (7) — MS relapse not requiring hospitalization

LIMITATIONS AND CAVEATS:
The study's nature required long waiting periods for pregnancies, and not all pregnant pwMS were open to enrollment. The demands of early motherhood led to significant drop-out rates over the four follow-up visits. Many patients opted out of starting natalizumab post-delivery as initially intended. These factors, combined with the COVID-19 pandemic, which significantly impacted research participation, resulted in a small sample size and diminishing cases throughout the follow-up period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT03046251/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT03046251/ICF_001.pdf